CLINICAL TRIAL: NCT03933709
Title: CONTROLLED, RANDOMIZED, BLIND CLINICAL TRIAL OF EFFECT OF A NUTRITIONAL SUPPORT SYSTEM (DIET, SUPPLEMENTS AND PROBIOTIC) FOR IMPROVING GROSS MOTOR FUNCTION IN CEREBRAL PALSY
Brief Title: Effect of a Nutritional Support System for Improving Gross Motor Function in Cerebral Palsy
Acronym: ENSSIGMCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anahuac University (Other)
Responsible Party: Principal Investigator, Fernando Leal-Martinez, Principal Investigator, Anahuac University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014/03001
Record Dates: First submitted 2019-03-20; First posted 2019-05-01 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Nutrition Disorder, Child; Gross Motor Development Delay; Neuro: Cerebral Palsy; Diet Modification; Probiotics
MeSH Terms: conditions — Child Nutrition Disorders | interventions — Crisis Intervention

STUDY DESIGN:
Intervention Model Description: Exploratory Study
Who Masked: Outcomes Assessor
Masking Description: Throughout the study, the physical therapy given was the same for the three groups and was applied by CRIT therapists. These staff members were not involved in the protocol. The evaluators did not have access to any information about the treatment given to each child, and this ensured the blind part to the study was met.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Follow-up Group (FG) (No Intervention): dietary surveillance and conventional therapy
- Control Group (CG) (Active Comparator): deworming and WHO diet
  Interventions: Other: deworming; Other: recommended diet
- Intervention Group (IG) (Experimental): deworming and the Nutritional Support System (NSS)
  Interventions: Dietary Supplement: Nutritional Support System (NSS); Other: deworming

INTERVENTIONS:
Dietary Supplement: Nutritional Support System (NSS) — Envelope 1 4.9g of Spirulina, 100mg ascorbic acid, 5mg folic acid and 10mg of glutamine. Was to be added to shake 1 during the first 10 days. Envelope 2 1g PUFAs n-3 and was to be added to shake 2 which was given throughout the intervention. Envelope 3 4.9g of Spirulina Maximum, 100mg ascorbic acid, 5mg folic acid, 5.2g vegetable protein, 125mg nicotinic acid, 50mg zinc, 100 mcg selenium and 800 UI cholecalciferol. Was to be added to shake 1 from day 11 until the end of week 6, after which it was suspended for 10 days and substituted for envelope 5 and then to be retaken until the end of the intervention. Envelope 4. 1g arginine and was to be added to shake 3 from day 8 until the end of the intervention. Envelope 5 contained the same ingredients as envelope 3 with an additional 10mg glutamine and was to be added to shake 1 from the start of week 7 for 10 days, after which envelope 3 was restarted. Probiotic at a dosage of 200 mg every 12 hours for 3 days at the beginning and week 6
  Other Names: Intervention treatment
  Arms: Intervention Group (IG)
Other: deworming — nitazoxanide at a dosage of 7.5 mg / kg every 12 hours for 3 days.
  Arms: Control Group (CG); Intervention Group (IG)
Other: recommended diet — WHO Diet
  Arms: Control Group (CG)

SUMMARY:
Background: Most patients with cerebral palsy (CP) are dependent on parents due to the spasticity and limitations in their gross motor function. Additionally, many of them do not respond to physical therapy due to deterioration in their nutritional status, which is secondary to gastrointestinal disorders, parasitosis, dysbiosis and the catabolic state of the disease itself. Evidence suggests that greater independence and better clinical response can be achieved by correcting the nutritional status. However, basic treatments only contemplate the calculation of energy requirements and do not consider important nutrients in particular, supplementation with glutamine, arginine, zinc, selenium, colecalciferol, nicotinic acid, spirulina, omega 3, ascorbic acid, vegetal protein or even probiotics.

Objective: To determine the effect of using a nutritional support system (NSS) diet, supplements and probiotic on the gross motor function in children with CP with spastic diparesic and Gross Motor Function Classification System III (GMFCS III).

Material and methods: In an exploratory study with controlled clinical trial design, 30 patients were randomly assigned to receive: 1) dietary surveillance and conventional therapy (FG), 2) deworming and WHO diet (CG), or 3) deworming and the NSS (IG). The patients were recruited from the Children´s Telethon Rehabilitation Center (CRIT) in Tlalnepantla Estado de México. Males and females aged 4-12 years were included with CP and spastic diparesic GMFCS III, who had a full-time caregiver and whose parents agreed to participate. They were studied for thirteen weeks. Gross motor function was evaluated at baseline and at 7 and 13 weeks after therapy using the GMFM scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CP with spastic diparesia and GMFCS III
* Re-entry
* Presence and support of a full-time caregiver
* To tolerate oral feeding
* Parents or guardians agree in writing to participate in the project
* Patients treated at the CRIT of Tlalnepantla Edo. Mex
* That the children, in the case of being able to write, accept in writing to participate in the project

Exclusion Criteria:

* Presence of any other catabolic disease, which further increases the risk of malnutrition (renal, cardiovascular, pulmonary, hepatic, immunological)
* Have had infectious problems or have received antibiotic treatment 15 days prior to the start of the study.
* Have received botulinum toxin therapy in the last 4 months
* Muscle relaxants in the last 6 months
* Severe gastroesophageal reflux
* Patients with any type of surgery performed with a period shorter than 9 months
* That can walk by themselves

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2015-01-12 (Actual); Primary Completion 2015-12-18 (Actual); Study Completion 2017-04-07 (Actual)

PRIMARY OUTCOMES:
Change from Gross Motor function Measure at 7 and 13 weeks | The GMFM scale was performed at baseline time and weeks 7 and 13 after intervention.
  This scale assesses five general parameters:
  1. Lying (decubitus) and rolling over (GMFAV),
  2. Sitting (GMFB),
  3. Crawling and kneeling (GMFC),
  4. Standing (GMFD),
  5. Walking (GMFE) and one final total item (GMFF).
  The scoring system consists of 88 items and each one is valued based on the following criteria:
  0= No,
  1. start,
  2. Partially Complete,
  3. Complete, NE= Not evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Leal, Study Director — Universidad Anáhuac Norte

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-03-28): https://cdn.clinicaltrials.gov/large-docs/09/NCT03933709/Prot_SAP_000.pdf
  • Informed Consent Form (2014-03-28): https://cdn.clinicaltrials.gov/large-docs/09/NCT03933709/ICF_001.pdf